CLINICAL TRIAL: NCT02184741
Title: A Double-Blind, Randomized, Placebo-Controlled Study of GB-0998 in Patients With Unexplained Recurrent Miscarriage.
Brief Title: A Study of the Efficacy and Safety of GB-0998 in Patients With Unexplained Recurrent Miscarriage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Blood Products Organization (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B211-11
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2022-01-28 (Actual); Status verified 2021-10

CONDITIONS: Recurrent Miscarriage
Keywords: IVIG; Unexplained Recurrent miscarriage; Primary Recurrent miscarriage; Intravenous immunoglobulin
MeSH Terms: conditions — Abortion, Habitual | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Infusion of normal saline
  Interventions: Drug: Placebo
- GB-0998 (Experimental): Infusion of GB-0998 (Immunoglobulin)
  Interventions: Drug: GB-0998

INTERVENTIONS:
Drug: GB-0998 — Subjects received GB-0998 at 400 mg/kg body weight once daily for 5 days until 6 weeks and 6 days of gestation after confirmation of the gestational sac by ultrasonography.
  Other Names: Intravenous Immunoglobulin （Venoglobulin®IH，2.5g/50ml）
  Arms: GB-0998
Drug: Placebo — Subjects received the same dose of saline as GB-0998 for 5 days after confirmation of the gestational sac by ultrasonography, up to 6 weeks and 6 days of gestation.
  Other Names: normal saline
  Arms: Placebo

SUMMARY:
The present survey was conducted to evaluate the efficacy and safety of GB-0998(immunoglobulin) in the treatment of unexplained recurrent miscarriage in comparison to placebo using a multicenter, double-blind, intergroup comparison method.

DETAILED DESCRIPTION:
Among the patients whose risk factors for recurrent miscarriage are unknown who repeatedly miscarry or patients who repeatedly miscarry despite treatment for risk factors, those who have never given birth and have had four or more miscarriages. Patients were assigned into two groups, GB-0998 or placebo, and received 8 ml/kg body weight of GB-0998 (400 mg/kg body weight) or placebo once a day for 5 days. The primary efficacy endpoint was ongoing pregnancy rate at 22 weeks of gestation (excluding miscarriages associated with fetal chromosomal abnormalities) and one of the secondary endpoint was live birth rate.

ELIGIBILITY:
Inclusion Criteria

1. Patients with primary recurrent miscarriage
2. Patients with a history of at least 4 miscarriages (not including biochemical pregnancy in the count of prior miscarriages)
3. Patients with any of the following risk factors for recurrent miscarriage

【Patients with unknown risk factors】 Patients with normal test results for each of the following risk factors who have experienced miscarriage of a fetus with normal chromosome karyotype

1. Abnormal uterine morphology
2. Thyroid dysfunction
3. Chromosome abnormality in the couple
4. Positive antiphospholipid antibody
5. Factor XII deficiency
6. Protein S deficiency
7. Protein C deficiency

【Patients determined to have risk factors】 Patients with the following risk factors who have experienced miscarriage of a fetus with normal chromosome karyotype despite receiving treatment for these factors

1. Abnormal uterine morphology (septate uterus): Patients who have undergone surgery
2. Thyroid dysfunction: Patients receiving medical treatment
3. Incidentally positive antiphospholipid antibody, factor XII deficiency, protein S deficiency, protein C deficiency:Patients receiving combination therapy with aspirin and heparin 4．Regardless of whether or not risk factors are present, patients should have experienced at least 1 a miscarriage of a fetus with normal chromosome karyotype 5．Patients below the age of 42 years at the time of obtaining informed consent 6．Patients who can be admitted for at least the period from the start date of administration of the study drug to the date of examination and assessment 1 week after the start of administration of the study drug 7．Patients who have given written informed consent to participate in this study

Exclusion Criteria:

1. Patients with chromosome abnormalities in themselves or their partners that are risk factors for recurrent miscarriage, patients with antiphospholipid syndrome, and patients with incidentally positive antiphospholipid antibody (when the latest test result is positive)
2. Patients in whom complications of diabetes mellitus or impaired glucose tolerance has been identified, but who have not received appropriate treatment for this condition
3. Patients who have received intravenous immunoglobulin therapy as treatment for recurrent miscarriage in the past
4. Patients with a history of stillbirth at 22 weeks of gestation or later
5. Patients receiving treatment for malignant tumor
6. Patients with a history of thromboembolism
7. Patients with a history of shock or hypersensitivity in response to the ingredients of this drug or patients with hereditary fructose intolerance
8. Patients who have been diagnosed with IgA deficiency in the past or patients who have a serum IgA level of <5 mg/dL at laboratory tests at registration
9. Patients who have received another study drug within the period of 12 weeks prior to informed consent or who are currently participating in another clinical trial
10. Patients who are unsuitable for this study for any other reason, in the opinion of a principal investigator or sub-investigators

Max Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 99 (Actual)
Dates: Start 2014-06-03 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate (excluding miscarriages associated with fetal chromosomal abnormalities) | At 22 weeks of gestation
  To evaluate the effectiveness of the drug in preventing miscarriages, we examined the ongoing pregnancy rate at 22 weeks and 0 days of gestation in cases excluding cases of fetal chromosome aberration miscarriages.

SECONDARY OUTCOMES:
Ongoing pregnancy rate(all patients) | At 22 weeks of gestation
  To evaluate the effectiveness of the drug in preventing miscarriages, we examined the ongoing pregnancy rate at 22 weeks and 0 days of gestation in all patients.
Live birth rate (excluding miscarriages associated with fetal chromosomal abnormalities) | At the time of birth
  To evaluate the effectiveness of the drug in total outcome of pregnancy, we examined the live birth rate in cases excluding cases of fetal chromosome aberration miscarriages.
Live birth rate(all patients) | At the time of birth
  To evaluate the effectiveness of the drug in total outcome of pregnancy, we examined the live birth rate in all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hideto Yamada, Director, Principal Investigator — Center for Recurrent Pregnancy Loss, Teine Keijinkai Hospital; Shigeru Saito, Professor, Principal Investigator — University of Toyama
Locations (1):
- Japan Blood Products Organization, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yamada H, Deguchi M, Saito S, Takeshita T, Mitsui M, Saito T, Nagamatsu T, Takakuwa K, Nakatsuka M, Yoneda S, Egashira K, Tachibana M, Matsubara K, Honda R, Fukui A, Tanaka K, Sengoku K, Endo T, Yata H. Intravenous immunoglobulin treatment in women with four or more recurrent pregnancy losses: A double-blind, randomised, placebo-controlled trial. EClinicalMedicine. 2022 Jun 29;50:101527. doi: 10.1016/j.eclinm.2022.101527. eCollection 2022 Aug. PMID 35795714